CLINICAL TRIAL: NCT03566355
Title: A Phase II Study of Curative Proton Beam Therapy for Patients With Lung Metastasis of Colorectal Cancer
Brief Title: Curative Proton Beam Therapy for Patients With Lung Metastasis of Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, DAE YONG KIM, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2018-0107
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer
Keywords: Lung Metastasis, Curative Proton Beam Therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- curative proton therapy (Experimental): Patients who meet the selection criteria are selected, signed for consent, and treated with proton therapy alone at 7200 cGy / 15 fractions, 5 times a week for 3 weeks
  Interventions: Radiation: curative proton therapy

INTERVENTIONS:
Radiation: curative proton therapy — Patients who meet the selection criteria are selected, signed for consent, and treated with proton therapy alone at 7200 cGy / 15 fractions, 5 times a week for 3 weeks

SUMMARY:
Proton alone therapy is performed

-> 5 times a week, 7200 cGy / 15 fractions for 3 weeks total

DETAILED DESCRIPTION:
This clinical trial is a prospective, single-organ, phase II clinical trial to evaluate the efficacy of curative proton therapy for pulmonary metastasis of colon cancer diagnosed histologically as adenocarcinoma.

Patients who meet the selection criteria should be selected, signed for consent, and treated 5 times a week for 7200 cGy / 15 fractions alone for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed colon adenocarcinoma in primary or metastatic lesions..
2. If there is no other remote metastasis other than lung, or if there is, control is possible
3. If there are less than 2 lung metastatic lesions
4. If they refuse lung surgery or surgery is inappropriate (medically unsuitable for surgery due to surgery refusal, diabetes mellitus, high blood pressure, pulmonary disease, heart disease, etc., repeated surgery, poor systematic function, short disease-free period, etc.)

Exclusion Criteria:

1. Other histologic cancer other than adenocarcinoma of the colorectal
2. Colorectal cancer without primary lesion resection
3. If there is another remote metastasis and is not completely resected or regulated
4. If the patient has experience of other invasive cancer diagnosis within 5 years of colorectal cancer diagnosis
5. Pregnancy and women under lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-05-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year local control ratio of the treated lung area | up to 3 years
  The primary goal of this study is the 3-year local control rate of pulmonary lesions treated with proton therapy. It is judged that the local control rate is improved when the pulmonary metastases of colorectal cancer using conventional X-ray is assumed to have 3-year local control rate of 60% and the 3-year local control rate of proton therapy is set to 80% or more

SECONDARY OUTCOMES:
3-year survival rate of treated patients | documented data of death, up to 3 years
  To evaluate whether high doses of proton therapy can replace conventional surgical resection. From date of initiation of proton therapy until the date of documented date of death from any cause, assessed up to 3 years
3-year disease-free survival rate of treated patients | documented date of progression or death, up to 3 years
  To evaluate whether high doses of proton therapy can replace conventional surgical resection. From date of initiation of proton therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Yong Kim, M.D., Principal Investigator — National Cancer Center Korea(South Korea)
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided